CLINICAL TRIAL: NCT02456584
Title: Pharmacodynamics (Suppression of Ovulation) and Pharmacokinetics Following a Single Subcutaneous Administration of Depo Provera® CI 150 mg/mL, Depo Provera® CI 300 mg/2 mL, or During Two Cycles of Depo-subQ Provera 104®
Brief Title: Pharmacodynamics and Pharmacokinetics Study of Existing DMPA Contraceptive Methods
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: FHI 360 (Other)
Collaborators: Oregon Health and Science University (Other); Asociación Dominicana Pro Bienestar de la Familia, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 702179
Record Dates: First submitted 2015-05-11; First posted 2015-05-28 (Estimated); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Contraception
Keywords: depot medroxyprogesterone acetate (DMPA); confidence interval (CI); Subcutaneous (sub-Q); Intrauterine device (IUD); Levonorgestrel (LNG); intrauterine system (IUS)
MeSH Terms: interventions — Injections, Intramuscular; Medroxyprogesterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- DMPA 150 (Experimental): single subcutaneous injection of 150mg/mL of DMPA in the abdomen
  Interventions: Drug: DMPA 150
- DMPA 300 (Experimental): single subcutaneous injection of 300mg/2mL of DMPA in the abdomen
  Interventions: Drug: DMPA 300
- DMPA 104 (Active Comparator): two injections, given at three months intervals, of 104mg/0.65mL of DMPA in the abdomen
  Interventions: Drug: DMPA 104

INTERVENTIONS:
Drug: DMPA 150 — injectable contraceptive
  Other Names: Depo-Provera® CI (150mg/mL, intramuscular)
  Arms: DMPA 150
Drug: DMPA 300 — injectable contraceptive
  Other Names: Depo-Provera® CI (300mg/2mL, intramuscular)
  Arms: DMPA 300
Drug: DMPA 104 — injectable contraceptive
  Other Names: depo-subQ provera 104® (104mg/0.65mL, sub-cutaneous)
  Arms: DMPA 104

SUMMARY:
This is a randomized, multi-center, parallel-group Phase I study to evaluate the pharmacodynamics (PD) of Medroxyprogesterone Acetate (MPA) after a single subcutaneous (SC) injection of 150 mg/mL or 300 mg/2 mL Depo-Provera CI in the abdomen of women of reproductive age with a confirmed ovulatory baseline cycle.

DETAILED DESCRIPTION:
This is a randomized, multi-center, parallel-group Phase I study with a primary objective to evaluate the pharmacodynamics (PD) of Medroxyprogesterone Acetate (MPA) after a single subcutaneous (SC) injection of 150mg/mL or 300mg/2mL Depo-Provera CI in the abdomen of women of reproductive age with a confirmed ovulatory baseline cycle.

Secondary study objectives are:

* To evaluate and compare the pharmacokinetics (PK) of MPA after a single SC injection of 150mg/mL or 300mg/2mL of Depo-Provera CI to two injections of Depo-subQ 104 administered 3 months apart
* To evaluate the relationship between serum MPA concentration and suppression of ovulation
* To evaluate and compare the safety, tolerability and acceptability of a SC injection of DMPA of different frequencies, doses and volumes

ELIGIBILITY:
inclusion

Women may be included in the study if they meet all of the following criteria:

* in good general health
* age 18 to 40 years, inclusive
* willing to provide informed consent and follow all study requirements
* not pregnant
* does not desire to become pregnant in the next 24 months
* regular menstrual cycle (24 to 35 days)
* confirmed ovulation by serum P ≥ 4.7 ng/mL in two consecutive samples during the pre-treatment phase of the study
* at low risk of pregnancy (e.g., sterilized, in exclusively same sex partnership, in monogamous relationship with vasectomized partner, abstinent, using non-hormonal IUD or condoms)
* has a body mass index of 18.0 to 35.0
* has hemoglobin ≥10.5 g/L

exclusion

Women will be excluded from participating in this study if they meet any of the following criteria:

* medical contraindications to DMPA use
* use of any of the following medications within 1 month prior to enrollment:

  * any investigational drug
  * prohibited drugs (per protocol)
  * oral contraceptives
  * LNG IUS or implant
* use of DMPA in the past 12 months
* use of a combined injectable contraceptive in the past 6 months
* recent pregnancy (within 3 months)
* current lactation
* ongoing or anticipated use of prohibited drugs (per protocol)
* known sensitivity to MPA
* plan to move to another location in the next 18 months
* any condition (social or medical) which in the opinion of the site investigator would make study participation unsafe, would interfere with adherence to study requirements or complicate data interpretation.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2015-09; Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Measure of time to ovulation | up to 18 months

SECONDARY OUTCOMES:
Cmax | up to 18 months
  Up to ovulation or 18 months following injection, whichever comes first
Aggregate of individual Cmax measurements and parameters | up to 18 months
Type and frequency of adverse events | up to 18 months
Blood pressure at follow up | up to 18 months
Pulse at follow up | up to 18 months
Weight at follow up | up to 18 months
Measure of delayed return to ovulation | up to 18 months
Serum concentrations of cortisol | 7.5 months
Number of participants with Injection site reactions | up to 18 months
Product acceptability | up to 18 months
Tmax | up to 18 months
  Up to ovulation or 18 months following injection, whichever comes first
Aggregate of individual Tmax measurements and parameters | Up to 18 months
MPA concentration at Day 91 (C91) | 91 days after injection
Aggregate of individual C91 measurements and parameters | 18 months after injection
MPA concentration at Day 182 (C182) | 182 days after injection
Aggregate of individual C182 measurements and parameters | 18 months after injection
MPA concentration at Day 210 (C210) | 210 days after injection
Aggregate of individual C210 measurements and parameters | 18 months after injection
Area under the curve (AUC 0-182) | 182 days after injection
Terminal elimination half-life (t1/2) | up to 18 months
  Up to ovulation or 18 months following injection, whichever comes first

CONTACTS AND LOCATIONS:
Overall Officials: Vera Halpern, MD, Study Director — FHI 360
Locations (2):
- Oregon Health & Science University, Portland, Oregon, United States
- Asociación Dominicana Pro Bienestar de la Familia, Inc. (PROFAMILIA), Santo Domingo, Dominican Republic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Halpern V, Brache V, Taylor D, Lendvay A, Cochon L, Jensen JT, Dorflinger LJ. Clinical trial to evaluate pharmacokinetics and pharmacodynamics of medroxyprogesterone acetate after subcutaneous administration of Depo-Provera. Fertil Steril. 2021 Apr;115(4):1035-1043. doi: 10.1016/j.fertnstert.2020.11.002. Epub 2021 Jan 21. PMID 33485608